CLINICAL TRIAL: NCT05428826
Title: Early Discontinuation of Steroid Treatment in Negative FDG-PET/CT Patients With Idiopathic Retroperitoneal Fibrosis. A Prospective Multicentric Study
Brief Title: Early Discontinuation of Steroid Treatment in Negative FDG-PET/CT Patients With Idiopathic Retroperitoneal Fibrosis
Acronym: METRO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP210082
Record Dates: First submitted 2022-06-07; First posted 2022-06-23 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Retroperitoneal Fibrosis
Keywords: Steroid treatment
MeSH Terms: conditions — Retroperitoneal Fibrosis | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Phase 4 Prednisone Dose : 1mg/kg/day at inclusion Route of administration : oral Duration of treatment: 9 to 21 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prednisone (Experimental): Dose : 1mg/kg/day at inclusion Route of administration : oral Duration of treatment: 9 to 21 months.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Phase 4 Prednisone Dose : 1mg/kg/day at inclusion Route of administration : oral Duration of treatment: 9 to 21 months.

SUMMARY:
Adult patients with a diagnosis of idiopathic retroperitoneal fibrosis Prospective multicentric cohort study Intervention : administration of prednisone during 9 to 21 months at 1mg/kg/day at inclusion.

DETAILED DESCRIPTION:
At baseline visit: Eligible patients will be screen during a standard visit care (consultation or hospitalization). A clinical examination, an abdominal CT scan, blood and urine biological tests will be performed.

At inclusion visit: After verification of inclusion and non inclusion criteria, if the patient meets the eligibility criteria, the investigator, will provide the patient with information and details regarding the trial. The consent is obtained and signed after a reflection period of 30 minutes.

The following procedure will be scheduled within 7 days:

* 18F-fluorodeoxyglucose-positron emission tomography (FDG-PET/CT) (pregnancy test if mandatory)
* Specimens for the biocollection Patients with positive FDG PET/CT (hypermetabolism grade II or III) at M0 will receive oral steroids (prednisone) at 1mg/kg/day during 1 month and then the dose will be tapered to obtain <10mg/day at 6 months and <7,5mg/day at 9 months.

Patients with a negative FDG-PET/CT (hypermetabolism grade 0 or I) at M0 will be excluded of the study.

Follow-up visits : M6, M9,M12,M15,M21, relapse At M6, M12, and M15: During these visits clinical examination (blood pressure measurement, body temperature, heart rate, weight and clinical signs or symptoms related to IRF) will be performed. An abdominal CT scan may be performed as part of the care depending on the clinician's judgment. Glucocorticoid compliance and tapering, concomitant medications and adverse events (including serious cardiovascular adverse events) will be assessed and recorded. A nurse will collect blood and urine.

At M9, M21 or relapse : During these visits clinical examination, an abdominal CT scan, a FDG-PET/CT blood and urine biological tests will be performed.

At M9: The patients who failed to reach remission at M9 are considered as treatment failure and will be treated on best medical judgment by the investigator and excluded to the study. The patients who had a dose of prednisone ≥7,5mg / day at M9 will also be excluded to the study.

Patients who achieved remission at M9 and have a retroperitoneal fibrosis visual score grade 0 or I under a dose of prednisone <7,5mg / day will discontinue steroids treatment.

Patients who achieved remission at M9 and have a retroperitoneal fibrosis visual score grade II or III under a dose of prednisone <7,5mg / day will continue steroids treatment at the actual dose (medical judgment).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* New onset or untreated relapsing of active idiopathic retroperitoneal fibrosis (IRF) defined by the association of:
* Related-disease symptoms (Appendix 17.2) or elevated CRP level (>20 mg/l) AND
* Retroperitoneal peri-aortic mass that surrounds the abdominal vessels on CT-scan

Exclusion Criteria:

* Secondary retroperitoneal fibrosis including drug-related retroperitoneal fibrosis, active infections (such as tuberculosis) or malignancies, systemic vasculitis (such as Anti-neutrophil cytoplasmic autoantibody (ANCA)-associated vasculitis), Erdheim-Chester disease (Appendix 17.3),patients with IgG4 disease may be enrolled
* Contraindication to perform FDG-PET/CT,
* Contraindication to perform CT scan with injection of contrast agent,
* Contraindication to treatment by prednisone
* Active infection
* Acute or chronic liver disease that is deemed sufficiently severe to impair their ability to participate in the trial,
* Active or history of malignancy in last 5 years. Individuals with squamous cell or basal cell skin carcinomas and individuals with cervical carcinoma in situ may be enrolled if they have received curative surgical treatment,
* Serum creatinine level greater than 400 µmol/L that cannot be attributed to underlying IRF,
* Live vaccination received from 4 weeks before inclusion,
* Inhaled glucocorticoids (except for patients with documented asthma),
* Any previous treatment with rituximab, methotrexate, alemtuzumab, cyclophosphamide, azathioprine, mycophenolate mofetil, infliximab, adalimumab, etanercept within the past 3 months,
* Pregnancy or breastfeeding,
* Non-affiliation to a social security regime,
* Subject deprived of freedom, subject under a legal protective measure
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2026-11-25 (Estimated); Study Completion 2028-11-25 (Estimated)

PRIMARY OUTCOMES:
To compare the cumulative IRF relapse rate 12 months after discontinuation of steroids. | 12 months after discontinuation of steroids
  The primary endpoint is the cumulate IRF relapse rate 12 months after discontinuation of steroids.
  The diagnosis of IRF relapse is based on the association of a clinical or biological criterion with a radiological criterion (i.e. composite criteria):
  * Clinical or biological criteria
    * recurrent or new-onset disease related symptoms
    * increase in C-reactive protein (CRP) >20mg/L without other cause
  * And a Radiological criterion o increased of retroperitoneal fibrosis size as compared with the CT scan performed at remission.
  The primary endpoint will be centrally adjudicated.

SECONDARY OUTCOMES:
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at inclusion | at inclusion
  Visual grades of retroperitoneal fibrosis FDG uptake as compared to liver FDG uptake (which consist of one item that yields a score of 0 to III),
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at inclusion | at inclusion
  maximal standardized uptake value (SUVmax) within the retroperitoneal fibrosis (regions of interest- ROI) at diagnosis (M0)
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at inclusion | at inclusion
  Metabolic volume (i.e. ratio of metabolically active volume (MAV) to global lesion volume) of retroperitoneal fibrosis FDG uptake at diagnosis
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at remission (M9) | 9 months after the inclusion
  Visual grades of retroperitoneal fibrosis fluorodeoxyglucose uptake as compared to liver fluorodeoxyglucose uptake (which consist of one item that yields a score of 0 to 3) A 0 significate an lack of FDG binding and a 3 an FDG uptake greater than liver uptakesignificate.
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at remission (M9) | 9 months after the inclusion
  maximal standardized uptake value (SUVmax) within the retroperitoneal fibrosis (regions of interest- ROI) at remission (M9)
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at remission (M9) | 9 months after the inclusion
  Metabolic volume (i.e. ratio of metabolically active volume (MAV) to global lesion volume) of retroperitoneal fibrosis FDG uptake remission (M9)
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at M21 | 21 months after the inclusion
  Visual grades of retroperitoneal fibrosis FDG uptake as compared to liver FDG uptake (which consist of one item that yields a score of 0 to III)
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at M21 | 21 months after the inclusion
  maximal standardized uptake value (SUVmax) within the retroperitoneal fibrosis (regions of interest- ROI) at M21
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at M21 | 21 months after the inclusion
  Metabolic volume (i.e. ratio of metabolically active volume (MAV) to global lesion volume) of retroperitoneal fibrosis FDG uptake at M21
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at relapse | between inclusion and 21 months after the inclusion
  Visual grades of retroperitoneal fibrosis FDG uptake as compared to liver FDG uptake (which consist of one item that yields a score of 0 to III)
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at relapse | between inclusion and 21 months after the inclusion
  maximal standardized uptake value (SUVmax) within the retroperitoneal fibrosis (regions of interest- ROI) at relapse
To analyze the characteristics of hypermetabolism of IRF in FDG-PET/CT and their evolution at relapse | between inclusion and 21 months after the inclusion
  Metabolic volume (i.e. ratio of metabolically active volume (MAV) to global lesion volume) of retroperitoneal fibrosis FDG uptake at relapse
To assess the performance of hypermetabolism of IRF in FDG-PET/CT for diagnosis of disease activity, | 21 months after the inclusion
  Diagnostic performance of SUVmax for the disease activity
To assess the performance of hypermetabolism of IRF in FDG-PET/CT for diagnosis of disease activity, | 21 months after the inclusion
  Diagnostic performance of MAV (area under the curve (AUC) and performance values for the Youden index) for the disease activity
To compare at M21 the corticosteroids therapy - related adverse events between patients who continue or discontinue the treatment at M9. | 21 months after the inclusion
  Frequency of diabetes, severe infection, osteoporotic fracture and major cardiovascular events 12 months after remission (M21). Serious cardiovascular adverse events are defined as a composite of nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death and will be assessed at M12,M15 and M21

CONTACTS AND LOCATIONS:
Overall Officials: Aline DECHANET, Study Chair — Assistance Publique - Hôpitaux de Paris (AP-HP)
Locations (15):
- France (15):
  - Médecine Interne, Agen, France
  - Médecine interne, Brest, France
  - Médecine interne et maladies infectieuses - GH Sud Haut Lévêque, Bordeaux
  - Médecine interne - Ambroise Paré, Boulogne-Billancourt
  - Médecine interne - Henri-Mondor, Créteil
  - Médecine interne et immunologie clinique - Dijon, Dijon
  - Médecine interne - Lille, Lille
  - Médecine Interne - La Timone, Marseille
  - Médecine interne - Saint Antoine, Paris
  - Médecine Interne, Vascularites et Myosites - La Pitié Salpêtrière, Paris
  - Médecine interne - Cochin, Paris
  - Médecine vasculaire - HEGP, Paris
  - Médecine Interne - Bichat, Paris
  - Néphrologie - Bichat, Paris
  - Médecine interne - Delafontaine, Saint-Denis

IPD SHARING:
Plan to Share IPD: No